CLINICAL TRIAL: NCT01414647
Title: The Effect of Diet Rich in Nordic Berries on Gut Microbiota, Glucose and Lipid Metabolism and Metabolism on Fenolic Compounds
Brief Title: The Health Effect of Diet Rich in Nordic Berries
Acronym: Berry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: VTT Technical Research Centre, Finland (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124//2005; 40361/05 (Other Grant/Funding Number: Tekes, National Technology Agency of Finland)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Syndrome; Impaired Glucose Tolerance; Low-grade Inflammation; Dyslipidemia
Keywords: Bilberry; Vaccinium myrtillus; Metabolic syndrome; Glucose metabolism; Lipid metabolism; Inflammation; Gene expression
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Dyslipidemias; Inflammation | interventions — Vaccinium myrtillus extract; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SRC (Experimental): Strawberry, raspberry and cloudberry intervention for 8 weeks
  Interventions: Dietary Supplement: 300 g of strawberry, raspberry and cloudberry
- BB (Experimental): Bilberry intervention for 8 weeks
  Interventions: Dietary Supplement: 400 g of bilberry
- C (Experimental): Control diet with restricted berry consumption
  Interventions: Other: Control diet

INTERVENTIONS:
Dietary Supplement: 300 g of strawberry, raspberry and cloudberry — 100 g of strawberry puree, 100 g of frozen raspberries and 100 g frozen cloudberries were concumed daily for 8 weeks. Bilberry consumption was restricted.
  Arms: SRC
Dietary Supplement: 400 g of bilberry — Equivalent amount to 400 g of fresh bilberries were consumed as 40 g of dried bilberries and as 200 g of frozen bilberries. Restriction of use of strawberries, raspberries and cloudberries were set.
  Arms: BB
Other: Control diet — Control diet, ie. habitual diet with restriction of berry consumption was consumed for eight weeks
  Other Names: Diet with restricted consumption of berries.
  Arms: C

SUMMARY:
Dietary polyphenols might have beneficial effects on glucose and lipid metabolism based on the studies made in animals or cell cultures. The findings regarding the possible decrease of low-grade inflammation are existing also in humans. Low-grade inflammation has been suggested to be a mechanistic link between obesity and its consequences on cardiometabolic health. The aim of the present study is to examine the effect of diet rich in berries on glucose and lipid metabolism and inflammatory markers.

DETAILED DESCRIPTION:
Berries are traditionally an important part of the Nordic diet. About 50 different berries are grown in the northern region, and about half of them are edible. Phenolic compounds are one of the most diverse group of secondary metabolites present in edible plants, and berries are especially rich in them. Flavonoids, phenolic acids, lignans and complex phenolic polymers (polymeric tannins) are typical for berries. Phenolic compounds are reported to have a variety of beneficial biological properties. They are potent antioxidants, and exhibit various other physiological activities including anti-inflammatory, antimicrobial, antiallergic, anticarcinogenic and antihypertensive activities. Epidemiological studies indicate that diet rich in phenolic compound correlates with lower risk of cancer and cardiovascular disease.

The aim of the present study is to examine the effect of diet rich in berries on glucose and lipid metabolism and inflammatory markers and gene expression profile in peripheral blood mononuclear cells (PBMCs) in subjects with features of metabolic syndrome.

Randomized, controlled clinical intervention including 4 wk run-in period, 8 wk dietary intervention and 4 wk recovery period was conducted.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI 26-39 kg/m2), and two of the following:
* elevated fasting plasma glucose in the absence of diabetes (5.6-6.9 mmol/l)
* abnormal serum lipid concentration: fasting serum triglyceride concentration >1.7 mmol/L, fasting serum HDL cholesterol <1.0 mmol/L (males) or <1.3 mmol/L (females))
* waist circumference >102 cm (males) or >88 cm (females)
* blood pressure >130/85 mmHg

Exclusion Criteria:

* chronic diseases
* use of lipid lowering medication

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Glucose level | week 8
  Fasting glucose level oral glucose tolerance status at study week 8
Cholesterol level | week 8
  total, HDL and LDL cholesterol level at the study week 8
Inflammation markers | week 8
  Various inflammation markers were measured at the study week 8

SECONDARY OUTCOMES:
Markers of sterol metabolism | week 8
  Markers of cholesterol absorption and synthesis were measured
gene expression in PBMCs | study week 8
  Global gene expression analyses in peripheral mononuclear cells (PBMC)

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Törrönen, Adjunct Professor, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Dpet of Public Health and Clinical Nutrition, Kuopio, Finland

REFERENCES:
- [Derived] Puupponen-Pimia R, Seppanen-Laakso T, Kankainen M, Maukonen J, Torronen R, Kolehmainen M, Leppanen T, Moilanen E, Nohynek L, Aura AM, Poutanen K, Tomas-Barberan FA, Espin JC, Oksman-Caldentey KM. Effects of ellagitannin-rich berries on blood lipids, gut microbiota, and urolithin production in human subjects with symptoms of metabolic syndrome. Mol Nutr Food Res. 2013 Dec;57(12):2258-63. doi: 10.1002/mnfr.201300280. Epub 2013 Aug 12. PMID 23934737
- [Derived] Kolehmainen M, Mykkanen O, Kirjavainen PV, Leppanen T, Moilanen E, Adriaens M, Laaksonen DE, Hallikainen M, Puupponen-Pimia R, Pulkkinen L, Mykkanen H, Gylling H, Poutanen K, Torronen R. Bilberries reduce low-grade inflammation in individuals with features of metabolic syndrome. Mol Nutr Food Res. 2012 Oct;56(10):1501-10. doi: 10.1002/mnfr.201200195. Epub 2012 Sep 7. PMID 22961907